CLINICAL TRIAL: NCT01213810
Title: Prevention of Varicella Zoster Virus (VZV)-Reactivation in HIV-positive Individuals Enrolled in a Prospective Immunogenicity and Safety Trial of VZV Vaccine: PROVE-IT-Study
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: SHCS 610
Record Dates: First submitted 2010-08-13; First posted 2010-10-04 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Herpes Zoster
Keywords: HIV; VZV (Varicella zoster Virus); vaccine; T cell; immunogenicity; safety
MeSH Terms: conditions — Herpes Zoster; Chickenpox | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Zostavax — Biological/Vaccine

SUMMARY:
The goal is to demonstrate the immunogenicity and safety of Zostavax® in HIV positive individuals. Study participants are stratified into different patient groups according to their CD4 cell count, viral load and HIV Status.

* Trial with medicinal product
* Trial with immunomodulatory product / biological

ELIGIBILITY:
Inclusion criteria: All individuals

* Age >18 years
* Male, or female with negative urine pregnancy test
* VZV-seropositive (serologically documented)
* Agree to use a barrier method of birth control (such as a condom)
* Written informed consent HIV positive individuals on ART (group A1-A3)
* Continuous ART for >3 months before baseline
* No change of ART regimen within 1 month before baseline
* HIV-RNA (value must be <3 months old )<50 copies/ml at last visit
* CD4-count (value must be <3 months old) > 500 cells/µl for group A1, 350-500 cells/µl for group A2 and 250 -349 cells/µl for group A3
* Participation in the SHCS HIV-positive individuals without ART (group B)
* HIV-1 RNA >1000 copies/ml (<3 months before baseline)
* CD4-cell count >500 cells/µl (<3 months before baseline)
* Participation in the SHCS Healthy HIV-negative volunteers (group C)
* Negative HIV-screening test (<3 months before baseline)
* CD4 cell count >500 cells/µl

Exclusion criteria: Common exclusion criteria

* Contraindications on ethical grounds
* Involvement in a conflicting (vaccine or investigational drug) clinical trial (except from the participation in the Swiss HIV Cohort Study).
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders or dementia of the subject.
* Pregnancy or breast feeding.
* Other clinically relevant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc),
* Known or suspected non-compliance, drug- or alcohol abuse.

Specific exclusion criteria

* Fever > 38.3 °C or acute illness during the last 4 weeks
* Exposure to chickenpox or shingles within four weeks prior to study entry
* History of shingles
* Immunosuppression due to disease (other than HIV) or due to medication within 30 days of study entry (eg corticosteroids)
* Household contact with known immunodeficiency (e.g. HIV-positive with CD4 <250 cells/µl)
* Immunoglobulin or blood product treatment within 1 year prior or 2 month after study vaccination
* Previous allergic reaction to vaccine components (i.e. neomycin or gelatin)
* Vaccination with a life attenuated vaccine one month prior to study entry
* History of chickenpox vaccination
* Treatment with anti-herpes drugs 4 weeks before baseline
* Severe coagulation disorder or oral anticoagulant treatment
* Laboratory exclusion criteria.

  * Thrombocytopenia < 50x 103/?l
  * Haemoglobin <12 g/dl
  * More than threefold elevation of ALT
  * Creatinine of more than150 µmol/l
  * Glucose >10 mmol/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity | half a year
  Geometric mean titer of Varicella zoster virus-specific IgG, VZV-specific T- cells per 106 peripheral mononuclear cells, Frequency of VZV-specific T- cells of total T-cells, CD4+ T-cells in different HIV-positive persons.
Safety | half a year
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability"

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Hasse, MD, Principal Investigator — University Hospital Zurich, Div of Infectious Diseases and Hospital Epidemiology